CLINICAL TRIAL: NCT07055776
Title: Compare the Effectiveness of Non-invasive Vagus Nerve Stimulation (nVNS) and Non-invasive Transcutaneous Electrical Nerve Stimulation (TENS) on Pain and Quality of Life (QOL) in Patients of Migraine: a Randomized Control Trial
Brief Title: Compare the Effectiveness of nVNS and TENS on Pain and Quality of Life in Patients of Migraine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/829
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-invasive vagus nerve stimulation (nVNS) (Experimental)
  Interventions: Combination Product: non-invasive vagus nerve stimulation (nVNS)
- non-invasive transcutaneous electrical nerve stimulation (TENS) (Experimental)
  Interventions: Combination Product: non-invasive transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Combination Product: non-invasive vagus nerve stimulation (nVNS) — Group 1 will receive non-invasive vagus nerve stimulation (nVNS) targeting the auricular branch of the vagus nerve (ABVN) using a TENS device with specialized ear clip electrodes. The electrodes will be placed on the cymba conchae or tragus region of the ear, where the ABVN is accessible. The stimulation parameters will be set to a frequency of 1 Hz (significantly reduced migraine headache), pulse width of 200-300 µs, and intensity adjusted to a strong but comfortable level without causing pain, applied for 15-30 minutes per session, 5 days a week for 12 weeks, based on protocols supported by evidence from studies such as Badran et al. (2018) and Yakunina et al. (2017), which demonstrated positive neuromodulatory effects through auricular stimulation. Baseline conventional physiotherapy for both groups will include: thermotherapy (e.g., moist hot packs for 15 minutes), range of motion (ROM) exercises, stretching of involved muscles, and strengthening exercises.
  Arms: non-invasive vagus nerve stimulation (nVNS)
Combination Product: non-invasive transcutaneous electrical nerve stimulation (TENS) — Group 2 will receive non-invasive transcutaneous electrical nerve stimulation (TENS) applied to the other areas to target other nerves stimulation (e.g., neck, upper trapezius, or occipital area). Surface electrodes will be placed paravertebrally, using a conventional TENS protocol: frequency of 20-25 Hz, pulse width of 200-300 µs, and intensity set to produce a strong but comfortable tingling sensation without muscle contraction. Each session will last 20-30 minutes, administered 5 days a week for 12 weeks. Baseline conventional physiotherapy for both groups will include: thermotherapy (e.g., moist hot packs for 15 minutes), range of motion (ROM) exercises, stretching of involved muscles, and strengthening exercises.
  Arms: non-invasive transcutaneous electrical nerve stimulation (TENS)

SUMMARY:
Migraine is a genetically influenced complex neurological disorder characterized by episodes of moderate-to-severe headaches, typically unilateral and frequently accompanied by nausea and heightened sensitivity to light and sound. The common type of migraine headaches is migraine without aura. Migraine has an approximate prevalence of 14.7%, making it the third most common disease in the world. This study aims to compare the effectiveness of non-invasive vagus nerve stimulation (nVNS) and non-invasive transcutaneous electrical nerve stimulation (TENS) in managing pain and improving quality of life (QOL) in patients with migraine.

ELIGIBILITY:
Inclusion Criteria:

* People will be eligible for participation of 18-75 years of age.
* Participants are included with previous diagnosis of migraine with aura according to ICHD-3 beta criteria.
* Patients who had 15 headache days per month over the last 6 months will be included in this study.

Exclusion Criteria:

* Participants with a history of secondary headaches,
* aneurysms, brain tumors, significant head trauma
* substance abuse, cardiovascular or cerebrovascular disease
* uncontrolled hypertension, psychiatric disorders,
* pregnancy, steroid use, botulinum toxin injections in the past 6 months, or certain other medical conditions were excluded.
* individuals with excessive use of pain medications, recent preventive treatments, or previous surgeries and procedures related to migraines will not be eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 12 Months
  The Visual Analogue Scale (VAS) is a simple tool used to measure the intensity of pain or symptoms. It typically uses a 10 cm (100 mm) horizontal line, where:
  0 = No pain 10 = Worst imaginable pain
HIT-6 (Headache impact test) | 12 Months
  The HIT-6 (Headache Impact Test) is a tool used to assess the impact of headaches, particularly migraines, on a person's daily life. It evaluates how headaches/pain affect daily functioning, work, social activities, and emotional well-being. The HIT-6 consists of 6 items. Each item is rated on a 5-point Likert scale (1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Very often, and 5 = Always). The individual responses are summed to obtain a total score that ranges from 36 to 78, with higher scores indicating greater headache impact and lower scores indicating less impact (below 50 suggests low impact, between 50 and 55 suggests moderate impact, and above 55 suggests severe impact).
MIDAS (Migraine Disability Assessment) | 12 Months
  The MIDAS (Migraine Disability Assessment) scale is a tool used to assess how migraines impact a person's daily life over the past three months. It includes five questions that ask about the number of days missed or affected in work, school, household tasks, and social activities due to migraines. The total number of days gives a MIDAS score, which is then categorized into four grades: Grade I (0-5) for little or no disability, Grade II (6-10) for mild, Grade III (11-20) for moderate, and Grade IV (21+) for severe disability. This helps clinicians evaluate the level of functional impairment caused by migraines

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No